CLINICAL TRIAL: NCT05143060
Title: Study on the Determination of Glycemic Index and Glycemic Load of Cereal Fiber Powder
Brief Title: Determination of Glycemic Index and Glycemic Load of Cereal Fiber Powder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: SYSEC-KY-KS-2020-203
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Glycemic Index
Keywords: Glycemic Index; Glycemic Load

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cereal fiber powder (Experimental): Cereal fiber powder
  Interventions: Dietary Supplement: Cereal powder
- Pure glucose powder (Placebo Comparator): Pure glucose powder
  Interventions: Dietary Supplement: Pure glucose powder

INTERVENTIONS:
Dietary Supplement: Cereal powder — Eat or drink oral glucose (reference) the valley of fiber powder upgrade formula, perfect meals, by extraction shu cereal bars, light appearance suits (by extraction shu compound dietary fiber powder, feeding combination 1:1) and 17 extraction enzyme 6 kinds of food respectively in different periods.
  Other Names: perfect meals; 17 extraction enzyme
  Arms: Cereal fiber powder
Dietary Supplement: Pure glucose powder — Pure glucose powder
  Arms: Pure glucose powder

SUMMARY:
This study choosed good health, aged 18 ~ 25, physical standard, the glucose tolerance test normal adults 12, oral glucose (reference) respectively in different periods, the valley of fiber powder upgrade formula, perfect meals, by extraction shu cereal bars, light appearance suits (by extraction shu compound dietary fiber powder, feeding combination 1:1) and 17 extraction enzyme 6 kinds of food, Venous blood was collected 15, 30, 45, 60, 90 and 120 min before and after oral administration respectively. Blood was collected for 7 times with 2mL each. The plasma is then separated to determine glucose levels. Blood glucose was measured within 3 h. With glucose as the reference, food glycemic index (GI) was calculated using the internationally used Wolever method. Time was taken as abscissa and blood glucose value at each time point was taken as ordinate to prepare the blood glucose response curve of each food tested after eating. The elevated glycemic area (AUC) under the glycemic curve was calculated geometrically, and the food GI and glycemic load (GL) values were calculated according to the following formula: GI value = (2 h post-meal blood glucose AUC of the tested food / 2 h post-meal glucose glucose AUC of the same amount of carbohydrate)×100, GL=GI*M(100g of the actual available carbohydrate of a food)/100.

DETAILED DESCRIPTION:
(I) Glucose test: twelve subjects began to fast at 10 PM the previous day, and 2mL of venous blood was collected on an empty stomach in the morning of the next day, which was divided into sodium fluoride anticoagulant tubes for measuring glucose. Then 25 g of pure glucose powder was taken orally, and venous blood was taken at 15, 30, 45, 60, 90 and 120 min, respectively. A total of 7 blood samples were collected, and 2mL of blood was collected each time. Then the plasma was separated to determine the content of glucose, and the blood glucose was measured within 3 h. In this study, venous indwelling needle was used to collect blood, which can reduce repeated venous aspiration. About 2 mL of normal saline was left in the indwelling needle to prevent blood clotting. Blood collection by an experienced nurse in charge or supervising nurse.

(II) Glucose response test of tested foods: Glucose test was conducted on the first day, and different tested foods (see Table 2 and Table 3) were tested on the third, sixth or ninth day respectively, with an interval of 2-3 days or more between the two foods. Specific dates were arranged according to the test schedule. Twelve subjects fasted after 10:00 PM the previous day, and 2mL of venous blood was taken on an empty stomach in the morning of the next day. They ate the tested food (containing about 25g or 10g carbohydrates, as shown in Table 2 and 3) on different dates respectively. The eating methods were as follows: The upgraded sample of grain fiber powder formula was washed and adjusted with 1:8 times of warm water at 60-70℃, stirred for about 2min and turned into a slightly thickened state, then put it at the palatability temperature and drink it. The perfect nutrition meal is rinsed with 1:6 times hot water at about 70℃, stirred evenly for about 1min, and then put it to the palatability temperature for drinking; Zhen Shu cereal bar pastry ready to eat in open bag; The nutritious meal + compound dietary fiber powder (good mixing according to the ratio of 1:1) is rinsed at 1:6 times in hot water around 70℃, stirred evenly for about 1min, and then put it to the palatability temperature for drinking; 17 light drink ferment drink directly after opening the bag. Venous blood was taken at 15, 30, 45, 60, 90 and 120 minutes, and blood glucose was measured within 3 hours. The blood collection method is the same as the above glucose test.

(3) Determination of plasma glucose: hexokinase method, with Beckman 5800 series automatic biochemical analyzer and its reagent determination.

(4) Calculation of food GI: With glucose as the reference (GI=100), the internationally used Wolever method was used to calculate food GI, with time as abscissa and blood sugar value at each time point as ordinate Postprandial glucose response curve. The elevated glucose area (AUC) under the glucose curve was calculated geometrically, and the food GI and GL values were calculated according to the following formula: GI value = (2 h post-meal blood glucose AUC of the tested food / 2 h post-meal glucose glucose AUC of the same amount of carbohydrate)×100, GL=GI*M(100g of the actual available carbohydrate of a food)/100.

(5) Quality control: (1) Formulate unified operation implementation methods and evaluation standards to standardize the operation; (2) Laboratory inspection requirements: unified methods, instruments and reagents; ③ Draw blood by experienced nurse in charge to ensure that the drawing time and indwelling needle meet the requirements; (4) Statistical processing and analysis methods of data were determined and implemented by statistical experts. Blood glucose quality control charts were drawn. Unified maximum allowable line and warning limit values were set according to the target value, and the measurement results should be within the warning line. ⑤ Set up inspectors to supervise the quality of each special work; ⑥ This study was in compliance with ethical standards, approved by the Ethics Committee of Sun Yat-sen Memorial Hospital of Sun Yat-sen University for filing, and informed consent signed by participating patients.

(VI) Data processing: The internationally used Wolever method was used to calculate the food GI. Using time as the abscissa and blood glucose values at each time point as the ordinate, the post-meal glucose response curves of the tested food were prepared and GI and GL were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, normal glucose tolerance test, normal blood pressure, no family history of diabetes or other metabolic history;
* Aged between 18 and 25;
* Normal body weight and waist circumference, body mass index (BMI) between 18.5 and 23.9kg/m2;
* No carbohydrate intolerance.

Exclusion Criteria:

* Those with abnormal glucose tolerance, overweight or obese, or lactose or carbohydrate intolerance were excluded.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Blood glucose was measured within 3 hours.
  Venous blood was collected up to 120 min

CONTACTS AND LOCATIONS:
Overall Officials: Chen C gang, Master, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Jenkins DJ, Wolever TM, Taylor RH, Barker H, Fielden H, Baldwin JM, Bowling AC, Newman HC, Jenkins AL, Goff DV. Glycemic index of foods: a physiological basis for carbohydrate exchange. Am J Clin Nutr. 1981 Mar;34(3):362-6. doi: 10.1093/ajcn/34.3.362. PMID 6259925
- [Background] Vrolix R, Mensink RP. Variability of the glycemic response to single food products in healthy subjects. Contemp Clin Trials. 2010 Jan;31(1):5-11. doi: 10.1016/j.cct.2009.08.001. Epub 2009 Sep 6. PMID 19737630
- [Background] Barclay AW, Petocz P, McMillan-Price J, Flood VM, Prvan T, Mitchell P, Brand-Miller JC. Glycemic index, glycemic load, and chronic disease risk--a meta-analysis of observational studies. Am J Clin Nutr. 2008 Mar;87(3):627-37. doi: 10.1093/ajcn/87.3.627. PMID 18326601